CLINICAL TRIAL: NCT05335551
Title: A Clinical Pilot Study to Test the Acceptability and Feasibility of TruGraf Liver and TRAC Liver Testing as Part of Standard of Care: Optimizing Liver ImmunoSuppression (TRU-IMMUNO)
Brief Title: TRU-IMMUNO: Optimizing Liver Immunosuppression
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Transplant Genomics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TGRP09
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Liver Transplant Rejection
Keywords: Biomarkers; Subclinical Rejection; Immunosuppression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients monitored with TruGraf/TRAC Liver testing: Subjects in the biomarker arm will have TruGraf Liver and TRAC Liver testing at study enrollment (1-2 months post-liver transplant) and thereafter every month for 6 months. Subjects will also have Trugraf Liver and TRAC Liver testing at months 9 and 12 following transplantation (7-8 and 10-11 months postbaseline)
  The TruGraf and TRAC Liver results will be used in the biomarker arm in conjunction with all other clinical parameters available to guide decisions of the Principal Investigator and Sub-Investigators related to immunosuppression management.
  changes.
  Interventions: Diagnostic Test: Patients monitored with TruGraf and TRAC Liver testing
- Patients not monitored with TruGraf/TRAC Liver testing: Patients in control/ stamdard of care arm will have immusuppresion reduction based on the clinical judgement and management of the Principal Investigator and Sub-Investigators.

INTERVENTIONS:
Diagnostic Test: Patients monitored with TruGraf and TRAC Liver testing — This is an observational study there are no protocol mandated interventions. TruGraf and TRAC Liver results will be utilized in conjunction with standard of care assessments to determine patient management in the study arm.
  Groups: Patients monitored with TruGraf/TRAC Liver testing

SUMMARY:
This is a prospective, multi-center, randomized study. The primary objective is to evaluate the feasibility and utility of TruGraf/TRAC Liver testing used in addition to standard of care measures of liver dysfunction to guide immunosuppression management.

DETAILED DESCRIPTION:
This study will provide TruGraf Liver and TRAC liver tests to one group of transplant providers early after liver transplantation to clarify if the Trugraf Liver and TRAC Liver results can complement their immunosuppression minimization strategies to avoid complications and reduce the occurrence of acute rejection. The ability to decrease IS will be compared to the group that does not receive the test results.

Subjects will be randomized into 2 groups: one will receive Trugraf/TRAC Liver testing and the other will not. Subjects in the biomarker arm will have TruGraf Liver and TRAC Liver testing at study enrollment (1-2 months post-liver transplant) and thereafter every month for 6 months. Subjects will also have Trugraf Liver and TRAC Liver testing at months 9 and 12 following transplantation (7-8 and 10-11 months post baseline). The TruGraf and TRAC Liver results will be used in the biomarker arm in conjunction with all other clinical parameters available to guide decisions related to immunosuppression changes. There are no protocol mandated immunosuppression changes. Subjects in the standard of care arm will not have biomarkers available for decisions related to immunosuppression changes.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Recipient of a primary or subsequent deceased-donor or living donor liver transplantation.
* Normal liver function tests at the time of or within 2 weeks of the baseline visit, defined by Total Bilirubin (TB) ≤1.5 mg/dL and Direct Bilirubin (DB) <0.5 mg/dL, Alkaline Phosphatase (AP) ≤200 U/L, and Alanine Transaminase (ALT) ≤60 U/L (males) ≤36 U/L (females).
* Between 1-2 months post-liver transplantation

Exclusion Criteria:

* Inability or unwillingness to provide informed consent.
* Recipients of previous hepatic or non-hepatic solid organ transplantation
* History of ≥2 mild or moderate rejections or 1 severe rejection prior to enrollment defined by BANFF 2016 criteria
* History of autoimmune liver disease
* Listed for repeat liver transplantation
* Infection with HIV
* Active HBV or HCV viremia (patients with undetectable virus can be included)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -This study is an observational study in adult (age ≥ 18 years), liver transplant patients who are 1-2 months post-transplantation. Approximately 130 subjects will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Immunosuppression reduction | 6-months
  Percent of subjects in each arm achieving at least 50% reduction from baseline total immunosuppressant (non-corticosteroid) dose at 6 months

SECONDARY OUTCOMES:
Immunosuppressant trough | 6-months
  Immunosuppressant trough levels at 6 months post transplant
Median and mean IS trough | 6-months
  Median and mean change in IS trough levels from baseline to 6 months
monotherapy immunosuppression | 1 year
  Percent of patients achieving monotherapy immunosuppression
clinical utility | 1 year
  Percent and total number of TruGraf Liver and TRAC Liver results that the PI identified as having clinical utility (Utility).
Liver testing workflow | 1 year
  Percent and total number of eligible patients for whom the PI was able to complete the entire TruGraf Liver and TRAC Liver testing workflow (Feasibility).
CKD score | 1 year
  Progression of CKD score managed by the KDIGO (Kidney Disease: Improving Global Outcomes) criteria from a scale of GI (normal kidney) to G5 (kidney failure)
BPAR for-cause biopsy | 1 year
  Incidence of biopsy proven acute rejection on a for cause biopsy at months 6 and 12
Acute rejection | 1 year
  Incidence of clinically treated acute rejection at months 6 and 12
eGFR timepoints | 1 year
  eGFR at months 6 and 12
eGFR timepoint range | 1 year
  eGFR change from baseline to months 6 and 12
Slope of eGFR | 1 year
  Slope of eGFR from baseline to months 6 and 12
eGFR decline or progression of CKD | 1 year
  Risk factors for eGFR decline or progression of CKD score
Infections | 1 year
  Incidence of grade 3 or greater infections at months 6 and 12
SF-36 scores | 1 year
  Change in SF-36 scores from baseline to 6 months and end of study (SF 36 is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Patty West-Thielke, PharmD, Principal Investigator — Transplant Genomics

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaked A, DesMarais MR, Kopetskie H, Feng S, Punch JD, Levitsky J, Reyes J, Klintmalm GB, Demetris AJ, Burrell BE, Priore A, Bridges ND, Sayre PH. Outcomes of immunosuppression minimization and withdrawal early after liver transplantation. Am J Transplant. 2019 May;19(5):1397-1409. doi: 10.1111/ajt.15205. Epub 2018 Dec 31. PMID 30506630
- [Background] Fischer L, Klempnauer J, Beckebaum S, Metselaar HJ, Neuhaus P, Schemmer P, Settmacher U, Heyne N, Clavien PA, Muehlbacher F, Morard I, Wolters H, Vogel W, Becker T, Sterneck M, Lehner F, Klein C, Kazemier G, Pascher A, Schmidt J, Rauchfuss F, Schnitzbauer A, Nadalin S, Hack M, Ladenburger S, Schlitt HJ. A randomized, controlled study to assess the conversion from calcineurin-inhibitors to everolimus after liver transplantation--PROTECT. Am J Transplant. 2012 Jul;12(7):1855-65. doi: 10.1111/j.1600-6143.2012.04049.x. Epub 2012 Apr 11. PMID 22494671
- [Background] Sterneck M, Kaiser GM, Heyne N, Richter N, Rauchfuss F, Pascher A, Schemmer P, Fischer L, Klein CG, Nadalin S, Lehner F, Settmacher U, Neuhaus P, Gotthardt D, Loss M, Ladenburger S, Paulus EM, Mertens M, Schlitt HJ. Everolimus and early calcineurin inhibitor withdrawal: 3-year results from a randomized trial in liver transplantation. Am J Transplant. 2014 Mar;14(3):701-10. doi: 10.1111/ajt.12615. Epub 2014 Feb 6. PMID 24502384
- [Background] Levitsky J, Asrani SK, Schiano T, Moss A, Chavin K, Miller C, Guo K, Zhao L, Kandpal M, Bridges N, Brown M, Armstrong B, Kurian S, Demetris AJ, Abecassis M; Clinical Trials in Organ Transplantation - 14 Consortium. Discovery and validation of a novel blood-based molecular biomarker of rejection following liver transplantation. Am J Transplant. 2020 Aug;20(8):2173-2183. doi: 10.1111/ajt.15953. Epub 2020 May 25. PMID 32356368
- [Background] Levitsky J, Kandpal M, Guo K, Zhao L, Kurian S, Whisenant T, Abecassis M. Prediction of Liver Transplant Rejection With a Biologically Relevant Gene Expression Signature. Transplantation. 2022 May 1;106(5):1004-1011. doi: 10.1097/TP.0000000000003895. Epub 2021 Jul 22. PMID 34342962
- [Background] Gielis EM, Ledeganck KJ, De Winter BY, Del Favero J, Bosmans JL, Claas FH, Abramowicz D, Eikmans M. Cell-Free DNA: An Upcoming Biomarker in Transplantation. Am J Transplant. 2015 Oct;15(10):2541-51. doi: 10.1111/ajt.13387. Epub 2015 Jul 16. PMID 26184824
- [Background] Sharon E, Shi H, Kharbanda S, Koh W, Martin LR, Khush KK, Valantine H, Pritchard JK, De Vlaminck I. Quantification of transplant-derived circulating cell-free DNA in absence of a donor genotype. PLoS Comput Biol. 2017 Aug 3;13(8):e1005629. doi: 10.1371/journal.pcbi.1005629. eCollection 2017 Aug. PMID 28771616
- [Background] Levitsky J, Kandpal M, Guo K, Kleiboeker S, Sinha R, Abecassis M. Donor-derived cell-free DNA levels predict graft injury in liver transplant recipients. Am J Transplant. 2022 Feb;22(2):532-540. doi: 10.1111/ajt.16835. Epub 2021 Sep 24. PMID 34510731
- [Result] Charlton M, Levitsky J, Aqel B, O'Grady J, Hemibach J, Rinella M, Fung J, Ghabril M, Thomason R, Burra P, Little EC, Berenguer M, Shaked A, Trotter J, Roberts J, Rodriguez-Davalos M, Rela M, Pomfret E, Heyrend C, Gallegos-Orozco J, Saliba F. International Liver Transplantation Society Consensus Statement on Immunosuppression in Liver Transplant Recipients. Transplantation. 2018 May;102(5):727-743. doi: 10.1097/TP.0000000000002147. PMID 29485508
- [Result] Levitsky J, O'Leary JG, Asrani S, Sharma P, Fung J, Wiseman A, Niemann CU. Protecting the Kidney in Liver Transplant Recipients: Practice-Based Recommendations From the American Society of Transplantation Liver and Intestine Community of Practice. Am J Transplant. 2016 Sep;16(9):2532-44. doi: 10.1111/ajt.13765. Epub 2016 Apr 22. PMID 26932352